CLINICAL TRIAL: NCT04349449
Title: A Prospective Observational Study of ENTYVIO Management in Crohn's Disease in Canada: Real-World Experience and Patient-Reported Outcomes
Brief Title: ENTYVIO in Bio-naive Patients With Moderate/Severe Crohn's Disease (CD) in Daily Practice
Acronym: EARLY-CD
Status: Withdrawn | Type: Observational
Why Stopped: Business Decision (no enrollment)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4022; U1111-1217-6862 (Registry Identifier: WHO); MACS-2017-102118 (Other: Study ID)
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vedolizumab Participants: Participants diagnosed with moderate to severe CD from approximately 20 investigational sites will be observed over a period of 12 months after initiation of treatment with vedolizumab, intravenous infusion under standard clinical care.

SUMMARY:
The purpose of this study is to describe physician-reported clinical effectiveness outcomes, as determined by Harvey-Bradshaw Index (HBI) assessment, in biologic-naive participants with CD over 12 months following treatment initiation with vedolizumab.

DETAILED DESCRIPTION:
This is a non-interventional, single-cohort, prospective study of participants with moderate to severe CD. The study will review medical charts with prospective patient-reported outcome measures to provide real-world data to describe clinical outcomes and participant-reported symptom experience over 12 months following vedolizumab treatment initiation.

The study will enroll approximately 140 participants. All participants will be enrolled in one observational group:

• Vedolizumab

This multicenter trial will be conducted in Canada. The overall duration of study will be approximately 24 months, including participant's enrolment period of 12 months and follow-up data collection period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Is enrolled in Takeda's participant support program prior to receiving vedolizumab.
2. Has a diagnosis of moderately-to-severely active CD, as documented in the medical records.
3. Scheduled for initial vedolizumab treatment per usual care recommendation.
4. Was biologic-naive at time of initiating vedolizumab treatment.

Exclusion Criteria:

1. Was prescribed vedolizumab as part of a clinical study.
2. Has isolated and active perianal disease in the absence of luminal CD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biologic-naive participants diagnosed with moderately to severely active CD who have initiated treatment with vedolizumab under standard clinical care will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants in Clinical Remission at Month 12 | Month 12
  Clinical remission is defined as HBI less than or equal to (<=) 5. HBI score is used to measure disease activity of CD. It consists of clinical parameters: general well-being (0= very well to 4= terrible), abdominal pain (0=none to 3= severe), number of liquid or soft stools/ previous day, abdominal mass (0= none to 3= definite and tender), and complications (8 items; 1 score/item). The total score is sum of sub scores, where score <5 = remission, 5 to 7 = mild disease activity, 8 to 16 = moderate disease activity and greater than (>) 16 = severe disease activity.

SECONDARY OUTCOMES:
Change From Baseline in HBI at Month 12 | Baseline up to Month 12
  HBI score is used to measure disease activity of CD. It consists of clinical parameters: general well-being (0= very well to 4= terrible), abdominal pain (0=none to 3= severe), number of liquid or soft stools/previous day, abdominal mass (0= none to 3= definite and tender), and complications (8 items; 1 score/item). The total score is sum of sub scores, where score <5 = remission, 5 to 7 = mild disease activity, 8 to 16 = moderate disease activity and >16 = severe disease activity.
Change From Baseline in Physician Global Assessment (PGA) at Month 12 | Baseline up to Month 12
  PGA score is used to measure disease activity of CD. Score ranges from 0 to 3, where 0 = normal condition; 1- mild disease condition; 2= moderate disease condition; and 3 = severe disease condition.
Change From Baseline in Patient-reported Outcome (PRO) Using the Two-item (PRO-2) at Month 12 | Baseline and Month 12
  The PRO2 is comprised of the stool frequency and abdominal pain components of the Crohn's Disease Activity Index (CDAI). The PRO-2 score is the sum of the abdominal pain and stool frequency subscores of the CDAI score. The average daily number of stools and abdominal pain score (with 0 indicating no pain and 4 indicating severe pain) over the past seven days are weighted according to the CDAI multiplication factors (2 for stool frequency and 5 for abdominal pain).
Change From Baseline in C-reactive Protein (CRP) Level at Month 12 | Baseline and Month 12
  Comparison of absolute change in CRP from baseline to Month 12. CRP is produced by the liver. The level of CRP rises when there is inflammation throughout the body.
Percentage of Participants in Remission as Determined by CRP Measurements <5 Milligram per Liter (mg/L) at Month 12 | Month 12
  Remission is defined as CRP <5 mg/L.
Change From Baseline in Fecal Calprotectin (FCP) Levels at Month 12 | Baseline and Month 12
Percentage of Participants in Remission as Determined by FCP Measurements (FCP < 50 milligram per kilogram [mg/Kg]) at Month 12 | Month 12
  Remission is defined as FCP <50 mg/kg.
Percentage of Participants With Endoscopic Improvement at Month 12 as Determined by Simple Endoscopic Score for Crohn's Disease (SES-CD) Values or Qualitative Physician Assessment of Disease Severity | Baseline and Month 12
  The SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and stenosis in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable is sum of values obtained for each segment. The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. The Physician's Assessment of Disease Severity was ranked on a 9-point scale (9 = much worse, 7 = worse, 5 = no change, 3 = better, 1 = much better).
Number of Participants Categorized by Participant Demographics, Clinical Characteristics and Disease Phenotype | Month 12
Change From Baseline in Work Productivity and Activity Impairment Specific Health Problem (WPAI-SHP) Score at Month 12 | Baseline, Month 12
  The WPAI-SHP assess the impact of CD on work productivity and daily activities, and classroom impairment during the previous 7 days. The questionnaire consists of questions about the number of hours missed from work, hours worked, and the extent to which work productivity and regular daily activities were affected. Scores will be calculated as percentages of hours worked and percentages of productivity at work on work days. An overall work productivity score will be computed by multiplying the percentage of work time by the percentage productivity at work; the higher the scores, the better work productivity and activity performance.
Change From Baseline in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Score at Month 12 | Baseline and Month 12
  The SIBDQ is a self-reported quantitative assessment of participant's health-related quality of life (HRQoL) in terms of physical, emotional, and social symptoms associated with IBD. The questionnaire relates to the past two weeks and consists of 10 questions about fatigue, social and leisure activities, pain, feelings of depression, and physical health issues. It consists of 7 point scale, with 1 indicating severity and 7 indicating the lack of a problem. The overall score can range from 10-70, with higher scores signifying better HRQoL.
Change From Baseline in Corticosteroid Dose at Month 12 | Baseline and Month 12
Change From Baseline in Immunomodulator Dose at Month 12 | Baseline and Month 12
Change From Baseline in the Percentage of Participants That are Steroid-free at Month 12 | Baseline and Month 12
Change From Baseline in the Percentage of Participants That are Immunomodulator-free at Month 12 | Baseline and Month 12
Number of Participants with Reporting one or More Adverse Events and Serious Adverse Events (SAEs) | Baseline up to Month 12
Number of Participants Based on CD-related Emergency Room (ER) Visits, Hospitalizations, or Surgeries | Baseline up to Month 12
Number of Participants that initiated Vedolizumab treatment and are still on Vedolizumab treatment at 12 months of follow-up | Baseline up to Month 12
Number of Participants With Reasons for Discontinuation of Vedolizumab Treatment | Baseline up to Month 12
Number of Participants Based on Subsequent Biologic Therapy Type | Baseline up to Month 12
Number of Participants that Received vedolizumab Dose Optimization | Baseline up to Month 12
  Dose optimization is defined as a change from every 8 weeks maintenance vedolizumab to any other schedule.
Time to vedolizumab Dose Optimization | Baseline up to Month 12
  Dose optimization is defined as a change from every 8 weeks maintenance vedolizumab to any other schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (14):
- Canada (14):
  - Kelowna GI Associates, Kelowna, British Columbia
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - The Winnipeg Clinic, Winnipeg, Manitoba
  - REGIONAL HEALTH AUTHORITY B doing business as HORIZON HEALTH NETWORK, Fredericton, New Brunswick
  - Nova ScotiaHealth Authority, Halifax, Nova Scotia
  - Barrie GI Associates, Barrie, Ontario
  - Lawson Health Research Institute a joint venture of London Health Science Centre Research Inc., Lawson Research Institute., London, Ontario
  - Girish Bajaj MPC, Oakville, Ontario
  - Sinai Health System, Toronto, Ontario
  - Kensington Cancer Screening Clinic, Toronto, Ontario
  - Toronto Immune and Digestive Health Institute, Toronto, Ontario
  - Research Institute McGill University Health Centre (RI-MUHC), Montreal, Quebec
  - Centre integre universitaire de sante et de services sociaux de l'Estrie Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.